CLINICAL TRIAL: NCT00112593
Title: Allogeneic Hematopoietic Stem Cell Transplantation for Induction of Mixed Hematopoietic Chimerism in Patients Infected With Human Immunodeficiency Virus-1 Using a Non-Marrow Ablative Conditioning Regimen Containing Total Body Irradiation in Combination With Post-Transplant Immunosuppression With Cyclosporine and Mycophenolate Mofetil
Brief Title: Fludarabine and Total-Body Irradiation Followed By Donor Stem Cell Transplant and Cyclosporine and Mycophenolate Mofetil in Treating HIV-Positive Patients With or Without Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ann Woolfrey, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1410.00; NCI-2010-00802 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1410.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); P01CA018029 (NIH); NCT00010348 (obsolete NCT alias)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Acute Undifferentiated Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Grade III Lymphomatoid Granulomatosis; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Aggressive NK-cell Leukemia; AIDS-related Diffuse Large Cell Lymphoma; AIDS-related Diffuse Mixed Cell Lymphoma; AIDS-related Diffuse Small Cleaved Cell Lymphoma; AIDS-related Immunoblastic Large Cell Lymphoma; AIDS-related Lymphoblastic Lymphoma; AIDS-related Peripheral/Systemic Lymphoma; AIDS-related Primary CNS Lymphoma; AIDS-related Small Noncleaved Cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Blastic Phase Chronic Myelogenous Leukemia; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Burkitt Lymphoma; Childhood Chronic Myelogenous Leukemia; Childhood Diffuse Large Cell Lymphoma; Childhood Grade III Lymphomatoid Granulomatosis; Childhood Immunoblastic Large Cell Lymphoma; Childhood Myelodysplastic Syndromes; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; Contiguous Stage II Adult Burkitt Lymphoma; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Contiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Contiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Contiguous Stage II Adult Lymphoblastic Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Essential Thrombocythemia; Extramedullary Plasmacytoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; HIV Infection; HIV-associated Hodgkin Lymphoma; Intraocular Lymphoma; Isolated Plasmacytoma of Bone; Juvenile Myelomonocytic Leukemia; Mast Cell Leukemia; Meningeal Chronic Myelogenous Leukemia; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Myeloid/NK-cell Acute Leukemia; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Polycythemia Vera; Post-transplant Lymphoproliferative Disorder; Previously Treated Myelodysplastic Syndromes; Primary Central Nervous System Lymphoma; Primary Myelofibrosis; Primary Systemic Amyloidosis; Progressive Hairy Cell Leukemia, Initial Treatment; Prolymphocytic Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage 0 Chronic Lymphocytic Leukemia; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Mixed Cell Lymphoma; Stage I Adult Diffuse Small Cleaved Cell Lymphoma; Stage I Adult Hodgkin Lymphoma; Stage I Adult Immunoblastic Large Cell Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Adult T-cell Leukemia/Lymphoma; Stage I Childhood Anaplastic Large Cell Lymphoma; Stage I Childhood Hodgkin Lymphoma; Stage I Childhood Large Cell Lymphoma; Stage I Childhood Lymphoblastic Lymphoma; Stage I Childhood Small Noncleaved Cell Lymphoma; Stage I Chronic Lymphocytic Leukemia; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Multiple Myeloma; Stage I Small Lymphocytic Lymphoma; Stage IA Mycosis Fungoides/Sezary Syndrome; Stage IB Mycosis Fungoides/Sezary Syndrome; Stage II Adult Hodgkin Lymphoma; Stage II Adult T-cell Leukemia/Lymphoma; Stage II Childhood Anaplastic Large Cell Lymphoma; Stage II Childhood Hodgkin Lymphoma; Stage II Childhood Large Cell Lymphoma; Stage II Childhood Lymphoblastic Lymphoma; Stage II Childhood Small Noncleaved Cell Lymphoma; Stage II Chronic Lymphocytic Leukemia; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma; Stage II Multiple Myeloma; Stage IIA Mycosis Fungoides/Sezary Syndrome; Stage IIB Mycosis Fungoides/Sezary Syndrome; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Childhood Anaplastic Large Cell Lymphoma; Stage III Childhood Hodgkin Lymphoma; Stage III Childhood Large Cell Lymphoma; Stage III Childhood Lymphoblastic Lymphoma; Stage III Childhood Small Noncleaved Cell Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage III Small Lymphocytic Lymphoma; Stage IIIA Mycosis Fungoides/Sezary Syndrome; Stage IIIB Mycosis Fungoides/Sezary Syndrome; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Childhood Anaplastic Large Cell Lymphoma; Stage IV Childhood Hodgkin Lymphoma; Stage IV Childhood Large Cell Lymphoma; Stage IV Childhood Lymphoblastic Lymphoma; Stage IV Childhood Small Noncleaved Cell Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Stage IVA Mycosis Fungoides/Sezary Syndrome; Stage IVB Mycosis Fungoides/Sezary Syndrome; T-cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
Keywords: HIV; Lymphoma; Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Lymphoma, Extranodal NK-T-Cell; Leukemia, Large Granular Lymphocytic; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Blast Crisis; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Thrombocythemia, Essential; HIV Infections; Intraocular Lymphoma; Leukemia, Myelomonocytic, Juvenile; Leukemia, Mast-Cell; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Polycythemia Vera; Primary Myelofibrosis; Immunoglobulin Light-chain Amyloidosis; Leukemia, Prolymphocytic; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Multiple Myeloma; Mycosis Fungoides; Sezary Syndrome; Waldenstrom Macroglobulinemia; Lymphoma; Leukemia | interventions — fludarabine phosphate; Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (allogeneic hematopoietic stem cell transplantation) (Experimental): CONDITIONING REGIMEN: Patients receive fludarabine IV over 2 hours on days -4, -3, and -2. Patients undergo TBI on day 0.
  TRANSPLANTATION: After completion of TBI, patients undergo allogeneic bone marrow or peripheral blood stem cell transplantation on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine IV or PO 2 to 3 times daily on days -3 to 99 with taper beginning on day 100 and continuing until day 177 in the absence of GVHD. Beginning within 6 hours after transplantation, patients also receive mycophenolate mofetil IV or PO 3 times daily on days 0 to 40 followed by a taper in the absence of GVHD.
  Interventions: Drug: fludarabine phosphate; Radiation: total-body irradiation; Procedure: peripheral blood stem cell transplantation; Drug: cyclosporine; Drug: mycophenolate mofetil; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Procedure: peripheral blood stem cell transplantation — Undergo allogeneic bone marrow or peripheral blood stem cell transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Drug: cyclosporine — Given IV or PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given IV or PO
  Other Names: Cellcept; MMF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies the side effects and best dose of giving fludarabine and total-body irradiation (TBI) together followed by a donor stem cell transplant and cyclosporine and mycophenolate mofetil in treating human immunodeficiency virus (HIV)-positive patients with or without cancer. Giving low doses of chemotherapy, such as fludarabine, and TBI before a donor bone marrow or peripheral blood stem cell transplant helps stop the growth of cancer or abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine (CSP) and mycophenolate mofetil (MMF) after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of treating high-risk HIV1-infected patients with 200 centigray (cGy) TBI plus post-transplant MMF/CSP.

II. To determine whether 200 cGy TBI plus post-transplant MMF/CSP results in stable mixed donor lymphocyte chimerism (5-95% donor cluster of differentiation [CD]3) in high-risk human immunodeficiency virus (HIV)-1 infected patients.

SECONDARY OBJECTIVES:

I. To define the kinetics of immune reconstitution following a non-lethal conditioning regimen in HIV1-infected patients.

II. To determine the effect of a non-lethal conditioning regimen on viral load.

OUTLINE:

CONDITIONING REGIMEN: Patients receive fludarabine intravenously (IV) over 2 hours on days -4, -3, and -2. Patients undergo TBI on day 0.

TRANSPLANTATION: After completion of TBI, patients undergo allogeneic bone marrow or peripheral blood stem cell transplantation on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine IV or orally (PO) 2 to 3 times daily on days -3 to 99 with taper beginning on day 100 and continuing until day 177 in the absence of graft-vs-host disease (GVHD). Beginning within 6 hours after transplantation, patients also receive mycophenolate mofetil IV or PO 3 times daily on days 0 to 40 followed by a taper in the absence of GVHD.

After completion of study treatment, patients are followed up for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancy, lymphoma or other HIV-associated malignancy are eligible provided these criteria are met:

  * The malignancy is in complete remission or very good partial remission, defined as a significant reduction of disease with therapy and no evidence for continued tumor growth in the case of lymphoma or solid tumors
  * Highly active antiretroviral therapy (HAART) is initiated within one month of hematopoietic cell transplant
  * Viral load has decreased by >= 1.5 logs or viral load < 5000 copies/ml plasma on HAART therapy
  * CD4 count is allowed to be > 100 cells/ul
* HIV infected patients without malignancy who have failed HAART are eligible provided that these criteria are met:

  * They have been treated with more than one regimen of HAART for a total of at least 6 months duration
  * The viral load is < 50 copies/ml plasma
  * The CD4 count < 100 cells/ul
* DONOR: Human leukocyte antigen (HLA) genotypically/phenotypically identical donor; if more than one HLA-identical sibling is available, priority will be given to donors matched for cytomegalovirus (CMV) status, ABO titer, and sex

  * Peripheral blood stem cells will be collected from donors greater than 12 years of age
  * Bone marrow will be collected from donors less than 12 years of age
* DONOR: HLA phenotypically identical unrelated donor; match grades allowed:

  * Match grade 1: Matched at allele level for HLA-A, B, C, DRB1, and DQB1
  * Match grade 2.1: Single allele disparity for HLA-A, B, C, DRB1, and DQB1

Exclusion Criteria:

* Positive serology for toxoplasma gondii on treatment or with evidence of active infection
* Patients with other disease or organ dysfunction that would limit survival to less than 30 days
* Patients with medical history of noncompliance with HAART or medical therapy
* DONOR: Donors for whom medical or psychologic reasons would make donor procedure intolerable
* DONOR: Marrow donors who have increased anesthetic risk
* DONOR: Donors who are HIV positive
* DONOR: Age > 75 years

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1999-11; Primary Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Woolfrey, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Woolfrey AE, Malhotra U, Harrington RD, McNevin J, Manley TJ, Riddell SR, Coombs RW, Appelbaum FR, Corey L, Storb R. Generation of HIV-1-specific CD8+ cell responses following allogeneic hematopoietic cell transplantation. Blood. 2008 Oct 15;112(8):3484-7. doi: 10.1182/blood-2008-05-157511. Epub 2008 Aug 12. PMID 18698002

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Allogeneic Hematopoietic Stem Cell Transplantation): CONDITIONING REGIMEN: Patients receive fludarabine IV over 2 hours on days -4, -3, and -2. Patients undergo TBI on day 0.
  TRANSPLANTATION: After completion of TBI, patients undergo allogeneic bone marrow or peripheral blood stem cell transplantation on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine IV or PO 2 to 3 times daily on days -3 to 99 with taper beginning on day 100 and continuing until day 177 in the absence of GVHD. Beginning within 6 hours after transplantation, patients also receive mycophenolate mofetil IV or PO 3 times daily on days 0 to 40 followed by a taper in the absence of GVHD.
  fludarabine phosphate: Given IV
  total-body irradiation: Undergo TBI
  peripheral blood stem cell transplantation: Undergo allogeneic bone marrow or peripheral blood stem cell transplantation
  cyclosporine: Given IV or PO
  mycophenolate mofetil: Given IV or PO
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Allogeneic Hematopoietic Stem Cell Transplantation)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Allogeneic Hematopoietic Stem Cell Transplantation)
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 43 [33 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Death From Regimen Toxicity or Opportunistic Infection
Time Frame: Within the first 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Hematopoietic Stem Cell Transplantation)
Number analyzed (Participants) | 5
Participants | 0

2. Primary Outcome: Death From GVHD
Time Frame: Within the first 360 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Hematopoietic Stem Cell Transplantation)
Number analyzed (Participants) | 5
Participants | 0

3. Primary Outcome: Successful Induction of Mixed Hematopoietic Chimerism as Assessed by the Percentage of Peripheral Blood T Cells That Are of Donor Origin
Description: Determined by a DNA-based assay that compares the profile of amplified fragment length polymorphisms (ampFLP) of the patient and donor.
Time Frame: Up to day 80
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Hematopoietic Stem Cell Transplantation)
Number analyzed (Participants) | 5
Participants | 5

4. Secondary Outcome: Overall Survival
Description: Kaplan-Meier estimate assessed at 1 year.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Treatment (Allogeneic Hematopoietic Stem Cell Transplantation)
Number analyzed (Participants) | 5
survival probability | 0.40 [0.14 to 1.00]

5. Secondary Outcome: Progression of HIV
Description: Count of participants with HIV progression.
Time Frame: Within 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Hematopoietic Stem Cell Transplantation)
Number analyzed (Participants) | 5
Participants | 0

6. Secondary Outcome: Reconstitution of HIV-specific Immunity
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic Hematopoietic Stem Cell Transplantation)
Number analyzed (Participants) | 4
Participants | 2

ADVERSE EVENTS:
Arm/Group | Treatment (Allogeneic Hematopoietic Stem Cell Transplantation)
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes